CLINICAL TRIAL: NCT00062062
Title: Parallel Phase II Trials of ZD1839 (Iressa) Alone or Weekly Carboplatin and Paclitaxel Followed by ZD1839 (Iressa) (Oncologists Must Choose) for Metastatic Non-Small Cell Lung Cancer in Patients > or = 65 Years of Age
Brief Title: Gefitinib With or Without Carboplatin and Paclitaxel in Treating Older Patients With Unresectable or Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0222; NCI-2012-02535 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000304453 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Lung Cancer
Keywords: stage IV non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Gefitinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- gefitinib (Experimental): Patients receive oral gefitinib on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Quality of life is assessed at baseline and after the completion of course 2.
  Patients are followed every 3 months for 5 years.
  Interventions: Drug: gefitinib
- paclitaxel + carboplatin + gefitinib (Experimental): Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. After completion of chemotherapy and in the absence of disease progression, patients receive oral gefitinib as in group I.
  Quality of life is assessed at baseline and after the completion of course 2.
  Patients are followed every 3 months for 5 years.
  Interventions: Drug: carboplatin; Drug: gefitinib; Drug: paclitaxel

INTERVENTIONS:
Drug: carboplatin
  Arms: paclitaxel + carboplatin + gefitinib
Drug: gefitinib
Drug: paclitaxel
  Arms: paclitaxel + carboplatin + gefitinib

SUMMARY:
RATIONALE: Biological therapies such as gefitinib may interfere with the growth of cancer cells and slow the growth of the tumor. Drugs used in chemotherapy such as carboplatin and paclitaxel use different ways to stop tumor cells from dividing so they stop growing or die. Combining gefitinib with carboplatin and paclitaxel may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gefitinib alone or together with carboplatin and paclitaxel works in treating older patients with unresectable or metastatic non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 6-month progression status of older patients with unresectable or metastatic non-small cell lung cancer treated with gefitinib alone or with carboplatin and paclitaxel.

Secondary

* Determine the response rate in patients treated with these regimens.
* Determine the quality of life of patients treated with these regimens.
* Determine whether serum-secreted or soluble epidermal growth factor receptor (EGFR) concentrations predict response in patients treated with these regimens.
* Correlate the presence of social support for these patients with toxicity and efficacy of these regimens.
* Determine whether social support for these patients differs according to gender.
* Determine the reasons an oncologist would choose a chemotherapy vs a nonchemotherapy regimen for these patients.

Tertiary

* Correlate EGFR signaling pathway markers, RNA expression profile, gene polymorphisms of prespecified germline and tumor genes, and plasma and urine proteomic patterns with response rate and time to progression of patients receiving treatment in group I.

OUTLINE: This is a nonrandomized, multicenter study. Patients are assigned to 1 of 2 treatment groups as determined by their treating physician.

* Group I: Patients receive oral gefitinib on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
* Group II: Patients receive paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. After completion of chemotherapy and in the absence of disease progression, patients receive oral gefitinib as in group I.

Quality of life is assessed at baseline and after the completion of course 2.

Patients are followed every 3 months for 5 years.

PROJECTED ACCRUAL: A total of 107 patients (51 for group I and 56 for group II) will be accrued for this study within 1.7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)

  * Metastatic or unresectable disease
* Measurable disease

  * At least 1 lesion at least 2.0 cm
  * Disease must be completely outside prior radiotherapy port OR documented disease progression since the completion of radiotherapy
* No meningeal carcinomatosis
* No untreated brain metastases

  * Current metastatic CNS disease must have been treated and clinically stable for at least 2 weeks prior to study chemotherapy
* No potentially curative treatment options available (e.g., chemotherapy with surgery or radiotherapy)

PATIENT CHARACTERISTICS:

Age

* 65 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10.0 g/dL

Hepatic

* Bilirubin no greater than 2.0 mg/dL
* No uncontrolled hepatic disease

Renal

* Creatinine no greater than 2 times upper limit of normal
* No uncontrolled renal disease

Cardiovascular

* No uncontrolled cardiac disease

Pulmonary

* No clinically active interstitial lung disease

  * Asymptomatic, chronic stable radiographic changes allowed
* No uncontrolled respiratory disease

Other

* Fertile patients must use effective contraception
* Able and willing to complete questionnaires alone or with assistance
* No known hypersensitivity to gefitinib or any of its excipients
* No active infection within the past 2 weeks
* No other prior malignancy within the past 5 years except basal cell skin cancer
* No grade 2 or greater peripheral neuropathy (CTC v2.0)
* No uncontrolled diabetes mellitus (for patients receiving study chemotherapy)
* No dysphagia or inability to swallow intact capsules
* No significant medical condition that would preclude study treatment or follow-up
* No severe or uncontrolled systemic disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No prior chemotherapy for metastatic NSCLC

Endocrine therapy

* Concurrent steroids allowed provided the dose is not changed

Radiotherapy

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered
* No prior radiotherapy to more than 25% of marrow-containing skeleton
* No concurrent radiotherapy (including palliative)

Surgery

* See Disease Characteristics
* At least 3 weeks since prior major surgery
* No surgery within 7 days after study participation

Other

* More than 30 days since prior non-FDA approved investigational drugs
* No concurrent oral retinoids
* No concurrent CYP3A4-inducing agents, including the following:

  * Carbamazepine
  * Oxcarbazepine
  * Modafinil
  * Ethosuximide
  * Griseofulvin
  * Nafcillin
  * Phenobarbital
  * Phenylbutazone
  * Phenytoin
  * Primidone
  * Rifampin
  * Hypericum perforatum (St. John's wort)
  * Barbiturates
  * Sulfinpyrazone
* No concurrent drugs that cause sustained elevation of gastric pH (≥ 5)
* No concurrent antacids within 4 hours before, during, and within 4 hours after gefitinib administration
* No concurrent itraconazole, fluconazole, ketoconazole, or erythromycin

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 65 (Actual)
Dates: Start 2004-10; Primary Completion 2006-08 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Progression status at 6 months | at 6 months

SECONDARY OUTCOMES:
Confirmed response rate (complete or partial response) | Up to 5 years
Overall survival | Up to 5 years
Progression-free survival | Up to 5 years
Quality of life as assessed by the Lung Cancer Symptom scale | Up to 5 years
Social support measure as assessed by the Lubben Social Network scale | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (141):
- United States (140):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - St. Anthony's Memorial Hospital, Effingham, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates at June E. Nylen Cancer Center, Sioux City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Cancer Center of Kansas, P.A. - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, P.A. - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, P.A. - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, P.A. - Newton, Newton, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, P.A. - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, P.A. - Salina, Salina, Kansas
  - Cancer Center of Kansas, P.A. - Wellington, Wellington, Kansas
  - Associates in Womens Health, P.A. - North Review, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, P.C., Lambertville, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Alexandria, Minnesota
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Brainerd Medical Center, Brainerd, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, P. C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Kenton Oncology, Incorporated, Kenton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Promedica Cancer Center at Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical College of Ohio Cancer Institute, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Toledo Surgical Specialists, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, P. C., Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Franciscan Skemp Healthcare, La Crosse, Wisconsin
- Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan, Canada

REFERENCES:
- [Result] Mc Kean H, Stella PJ, Hillman SL, Rowland KM, Cannon MW, Behrens RJ, Gross GG, Sborov MD, Friedman EL, Jatoi A. Exploring therapeutic decisions in elderly patients with non-small cell lung cancer: results and conclusions from North Central Cancer Treatment Group Study N0222. Cancer Invest. 2011 May;29(4):266-71. doi: 10.3109/07357907.2010.535061. Epub 2011 Feb 23. PMID 21345074